CLINICAL TRIAL: NCT01350258
Title: A Two Step Approach to Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation for Hematologic Malignancies Using Melphalan for T-Cell Tolerization
Brief Title: Bone Marrow Transplant Using a Reduced Intensity Regimen That is Given in Two Steps
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10D.535; 2010-40 (Other: CCRRC); JT 2173 (Other: JeffTrial Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Malignancies; Acute Leukemia; Myelodysplastic Syndromes (MDS) Other Than RA or RARS Subtypes; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Myeloma; Chronic Myelogenous (or Myeloid) Leukemia (CML) Resistant to STI Therapy
Keywords: allogeneic HSCT; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell; Leukemia | interventions — fludarabine; fludarabine phosphate; Thiotepa; Whole-Body Irradiation; Radiotherapy; Melphalan; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant Treatment Group (Experimental): All patients treated on this research study.
  Interventions: Drug: Fludarabine; Drug: Thiotepa; Radiation: Total Body Irradiation (TBI); Biological: Donor Lymphocyte Infusion (DLI); Drug: Melphalan; Device: Hematopoietic stem cell transplantation (HSCT)

INTERVENTIONS:
Drug: Fludarabine — Part of the conditioning regimen
  Other Names: fludarabine phosphate; Fludara
Drug: Thiotepa — Part of the conditioning regimen
  Other Names: N,N'N'-triethylenethiophosphoramide
Radiation: Total Body Irradiation (TBI) — There is one fraction of total body irradiation (2Gy) as part of the conditioning regimen.
  Other Names: radiotherapy
Biological: Donor Lymphocyte Infusion (DLI) — Immediately following the conditioning regimen of fludarabine, thiotepa, and TBI, the patient receives a set dose of their donor's T cells (DLI), After the DLI, the donor's T cells will react with the remaining parts of the recipients immune system.
  Other Names: buffy coat fusion
Drug: Melphalan — Two days after the DLI, Melphalan will be given to eliminate the reacting T cells to avoid graft versus host disease. Non-activated T cells should not be affected by the Melphalan and remain to help fight infection.
  Other Names: MEL; Melphalan hydrochloride; Alkeran
Device: Hematopoietic stem cell transplantation (HSCT) — One day after the Melphalan ends, the patient will receive their donor's stem cells. This is the actual day of transplant.
  The CliniMACS® Plus Instrument will be used for the selection of human CD34+ hematopoietic stem and progenitor cells in human allogeneic hematopoietic stem cell transplantation.
  Other Names: CliniMACS

SUMMARY:
This is a research study involving the treatment of patients with hematological cancers with allogeneic (cells from a donor) hematopoietic stem cell transplant (HSCT). HSCT is often referred to as bone marrow transplant. Patients who are not expected to have long term survival after conventional therapy will undergo HSCT as a curative therapy after receiving front line therapy for their disease. This project is based on an HSCT approach that has been used at TJU since 2006 with the goal of optimizing this type of treatment further. In this new study, the investigators will substitute the chemotherapy agent, Melphalan (Mel), for cyclophosphamide (CY). Cyclophosphamide was used in the original trial. The research question is whether side effects are less using Mel and if donor T cells can be made tolerant to the recipient with the use of Mel. The proposed study is also more specific in terms of performance status and organ function entry criterion. The investigators observed in the original trial that patients with poor performance upon admission for transplant did not have as good outcomes.

Because many older patients are treated according to this type of transplant, the chemotherapy and radiation used are less intensive than other types of transplant. The name for this in the transplant field is a reduced intensity hematopoietic stem cell transplant. The abbreviations most used in this document are RIC for reduced intensity conditioning, HSCT which refers to the transplant itself, and MEL which refers to the drug, Melphalan.

DETAILED DESCRIPTION:
Twenty-nine patients in the Thomas Jefferson University (TJU) Blood and Marrow Transplantation Program have been treated on the research protocol, A Two Step Approach To Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation for Hematologic Malignancies from HLA Partially-Matched Related Donors (TJU 2 Step RIC, TJU IRB# 06U.328) as of July, 2010. While treatment on this protocol has resulted in durable responses for many older patients and younger, heavily pretreated patients with hematological malignancies, poor performance status at the time of transplant and morbidities related to cyclophosphamide (CY) administration in the regimen have contributed to decreased survival. In addition, disease relapse after hematopoietic stem cell transplantation (HSCT) has been a major cause of mortality for those patients with disease at the time of transplant.

The objective of this research is to improve patient outcomes after treatment on the TJU 2 Step RIC protocol by refining the approach based on outcomes observed in the initial trial. More thorough assessment of performance status prior to HSCT and the substitution of the alkylating agent Melphalan (MEL) for CY to decrease CY-related toxicity while strengthening the anti-leukemic intensity of the regimen for patients with poor-risk disease will be the major strategies used to increase the efficacy of the regimen. MEL has shown efficacy against myeloid malignancies when used in conditioning in RIC HSCT. Patients with AML and MDS were the most common group treated on the initial TJU 2 Step RIC trial and also comprise the largest patient group treated in the TJU Medical Oncology Program.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a high-risk hematologic or oncologic diagnosis in which allogeneic HSCT is thought to be beneficial, and in whom front-line therapy has already been applied. High risk is defined as:

   * Acute leukemia in 3rd or greater CR or with persistent disease
   * Myelodysplastic syndrome (MDS) other than RA or RARS subtypes.
   * Hodgkin's or Non-Hodgkin's lymphoma in 3rd or greater remission or with persistent disease.
   * Myeloma in 3rd or greater remission or with less than PR to most recent therapy.
   * Chronic myelogenous (or myeloid) leukemia (CML) resistant to STI therapy
2. Patients must have a related donor who is at least a 4 antigen match at the HLA-A; B; C; DR loci.
3. Patients must adequate organ function:

   * LVEF of > or = 50%
   * DLCO > or = 50% of predicted corrected for hemoglobin
   * Adequate liver function as defined by a serum bilirubin < or = 1.8, AST or ALT < or = 2.5X upper limit of normal
   * GFR of > or = 60 mL/min/1.73m2
4. Performance status > or = 80% (TJU Karnofsky) for patients > or = 60 years old or > or = 70% for patients < 60.
5. HCT-CI Score < or = 4 points for patients > or = 60 years old or < or = 5 points for patients < 60.
6. Patients must be willing to use contraception if they have childbearing potential
7. Able to give informed consent

Exclusion Criteria:

1. Performance status < 80% (TJU Karnofsky) for patients > or = 60 years old or < 70% for patients < 60.
2. HCT-CI Score > 4 points for patients > or = 60 years old or > 5 points for patients < 60.
3. HIV positive
4. Active involvement of the central nervous system with malignancy
5. Inability to obtain informed consent
6. Pregnancy
7. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder
8. Patients who have received alemtuzumab within 8 weeks of the transplant admission, or who have recently received horse or rabbit ant-thymocyte globulin and have an ATG level of > or = 2 ugm/ml
9. Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol

Donor Selection All donors are selected and screened for their ability to provide adequate infection-free apheresis products for the patient in a manner that does not put the donor at risk for negative consequences. Donor selection will be in compliance with 21 CFR 1271 and TJU BMT Program SOP CP: P009.03.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University; Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant Treatment Group: REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV over 60 minutes on days -11 to -8 and thiotepa IV (cytarabine IV as of February 2012) over 2 hours on days -11 to -9. Patients undergo TBI on day -6. Patients receive melphalan IV over 20 minutes on days -3 and -2.
  TRANSPLANTATION: Patients undergo DLI on day -6 and allogeneic CD-34+ peripheral blood stem cell transplantation on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO beginning on day -1 with taper beginning on day 42 and receive MMF IV BID on days -1 to day 28.
Period: Overall Study
Arm/Group | Transplant Treatment Group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.43 (7.86)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Defined Dose of Melphalan (MEL)
Description: To define the dose of MEL required for the establishment of peripheral T cell tolerance with concomitant immune reconstitution.
Time Frame: 100 days post-transplant
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 2: Non-Relapse Mortality (NRM)
Description: To evaluate the 100 day non-relapse mortality (NRM) rate in patients undergoing HSCT treated on this successor TJU 2 Step RIC haploidentical regimen and compare it with that of the initial regimen.
Time Frame: 100 days post-treatment
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Relapse Rate
Description: To compare relapse rates in patients undergoing HSCT treated on this successor TJU 2 Step RIC haploidentical regimen and compare it with that of the initial regimen.
Time Frame: At 1 and 3 years
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 0

4. Secondary Outcome: GVHD Incidence and Severity
Description: To determine the incidence and severity of graft-versus-host disease (GVHD) in patients undergoing treatment on this regimen using MEL for T cell tolerization as well as tacrolimus and mycophenolate mofetil (MMF) as GVHD prophylaxis.
Time Frame: At 1 and 3 years
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 0

5. Secondary Outcome: Engraftment Rate and Lymphoid Reconstitution
Description: To evaluate engraftment rates and lymphoid reconstitution in patients treated on this trial.
Time Frame: 100 days post-transplant
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: To assess overall survival in patients undergoing HSCT treated on this trial.
Time Frame: At 1 and 3 years
Arm/Group | Transplant Treatment Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Transplant Treatment Group
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Treatment Group (N=8)
CMV reactivation (Immune system disorders) | 2 (2)
Colitis/enteritis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Fever (General disorders) | 2 (2)
Gram negative sepsis (Blood and lymphatic system disorders) | 1 (1)
HHV-6 viremia (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 2 (2)
Hypoxia (General disorders) | 1 (1)
Increased LFTs (Hepatobiliary disorders) | 1 (1)
Lacunar infarct in pons (General disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
Orthostatic hypotension (Blood and lymphatic system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Treatment Group (N=8)
Abdominal cramping (General disorders) | 1 (1)
Abdominal pain (General disorders) | 6 (7)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1)
Anorexia (General disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 7 (7)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Back pain (General disorders) | 2 (2)
Balance problems (General disorders) | 1 (1)
Blister at PICC site (Skin and subcutaneous tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood in stool (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Body aches (General disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Buttocks wound (General disorders) | 1 (1)
Changes in vision (Eye disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
CMV reactivation (Immune system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Decreased appetite (General disorders) | 1 (2)
Decreased urine output (Renal and urinary disorders) | 2 (3)
Dehydration (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (10)
Disturbing dreams (Psychiatric disorders) | 1 (1)
Dizziness (General disorders) | 2 (2)
Dry eyes (Eye disorders) | 1 (1)
Dry mouth (General disorders) | 2 (4)
Dry nose/sinuses (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear fullness (Ear and labyrinth disorders) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 3 (3)
Electrolyte imbalance (General disorders) | 2 (2)
Increased LFTs (Hepatobiliary disorders) | 2 (3)
Erythematous mucosa in duodenal bulb (Gastrointestinal disorders) | 1 (1)
Eye movement abnormality (Eye disorders) | 1 (1)
Eye tearing (Eye disorders) | 1 (1)
Face/upper neck swelling (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Feels "fuzzy" (General disorders) | 1 (1)
Feet/ankle/leg swelling (General disorders) | 2 (3)
Fever (General disorders) | 7 (20)
Flank pain (General disorders) | 1 (1)
Fluid overload (Blood and lymphatic system disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Headache (General disorders) | 5 (8)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
HHV-6 viremia (Blood and lymphatic system disorders) | 2 (2)
Hiccups (General disorders) | 2 (3)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hypernatremia (Blood and lymphatic system disorders) | 3 (4)
Hyperphosphatemia (Blood and lymphatic system disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Blood and lymphatic system disorders) | 5 (5)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 3 (3)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 4 (4)
Hypothermia (General disorders) | 3 (4)
Hypoxia (General disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Increased creatinine (Blood and lymphatic system disorders) | 3 (3)
Insomnia (General disorders) | 3 (4)
Itchiness in throat (General disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Leg pain (General disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Mental status change (General disorders) | 5 (7)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 5 (5)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (General disorders) | 6 (8)
Neuropathy (Nervous system disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Non-productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Occult blood (Gastrointestinal disorders) | 2 (2)
Oral discomfort (General disorders) | 1 (1)
Orthostatic hypotension (Blood and lymphatic system disorders) | 2 (2)
Pain at PEG tube site (General disorders) | 1 (1)
Pericatheter thrombus (Blood and lymphatic system disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post nasal drip (General disorders) | 1 (1)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Ptosis (Eye disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Purulent drainage (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (12)
Renal failure (Renal and urinary disorders) | 2 (2)
Respiratory crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors/chills (General disorders) | 4 (4)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin tear (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (General disorders) | 2 (2)
Stomach fluttering (Gastrointestinal disorders) | 1 (1)
Sweats (General disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (6)
Tenderness at PICC site (General disorders) | 1 (1)
Thrush (Infections and infestations) | 2 (2)
Tingling in lips (General disorders) | 1 (1)
Tissue wound (Skin and subcutaneous tissue disorders) | 1 (1)
Tremors (General disorders) | 3 (3)
Trouble sleeping (General disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vision - flashing lights (General disorders) | 1 (1)
Vivid dreams/hallucinations (Psychiatric disorders) | 1 (1)
Volume overload (Cardiac disorders) | 3 (3)
Vomiting (General disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wrist tenderness (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to extreme toxicity. The study was closed before any data could be collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes